CLINICAL TRIAL: NCT05958550
Title: Construction and Validation of a Risk Prediction Model for Hypothermia After Laparoscopic Gastrointestinal Tumor Surgery Based on Machine Learning
Brief Title: A Risk Prediction Model for Hypothermia After Laparoscopic Gastrointestinal Tumor Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LY2023-072-B
Record Dates: First submitted 2023-06-06; First posted 2023-07-24 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Hypothermia; Anesthesia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypothermia group
  Interventions: Behavioral: The tympanic membrane temperature of patients was measured.
- Non-hypothermia group
  Interventions: Behavioral: The tympanic membrane temperature of patients was measured.

INTERVENTIONS:
Behavioral: The tympanic membrane temperature of patients was measured. — After the patient entered the anesthesia recovery room ( PACU ) at the end of the operation, the ear canal was cleaned with cotton swabs by nurses trained in the use of ear temperature guns to avoid the impact of earwax. The patient was in a supine position, the patient 's head was fixed, the patient 's auricle was gently pulled back and up, the ear canal was straight, the ear temperature gun was put into the ear canal, the temperature of the patient 's left and right ears was measured uniformly, and the average value was taken as the final body temperature value. Thereafter, the same measurement was performed every 20 minutes until the patient left the resuscitation room.

SUMMARY:
The incidence of postoperative hypothermia in patients with laparoscopic gastrointestinal tumors is high. Hypothermia increases the risk of postoperative complications and medical costs. Early warning can effectively reduce the incidence of postoperative hypothermia in patients. Multivariate prediction models help identify high-risk patients and reversible factors. At present, there are few reports on the risk factors and prediction models of postoperative hypothermia in patients with laparoscopic gastrointestinal tumors. Therefore, this study aims to clarify the risk factors of postoperative hypothermia in patients with laparoscopic gastrointestinal tumors. Four machine learning algorithms, traditional Logistic regression analysis, decision tree, random forest and naive Bayes, were used to establish risk prediction models. According to the TRIPOD statement, C-index, Hosmer-Lemeshow ( H-L ) test and decision curve analysis ( DCA ) were used to evaluate the prediction and fitting effects of the models in all aspects, and the optimal model was selected and verified. Provide reference for subsequent research.

ELIGIBILITY:
Inclusion Criteria:

* The types of surgery included laparoscopic radical gastrectomy for gastric cancer, duodenal cancer, colon cancer, rectal cancer and small bowel cancer. Age ≥ 18 years ; the anesthesia method was general anesthesia ; elective surgery.

Exclusion Criteria:

* Patients with abnormal body temperature such as fever and hypothermia before operation ; patients who need low temperature to protect organs during operation ; patients who were converted to laparotomy during the operation ; a clear diagnosis of sweat gland dysfunction ; patients with external auditory canal active disease ; reject participants.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: From June 2023 to January 2024, patients underwent laparoscopic gastrointestinal tumor surgery in the East Hospital of Renji Hospital, Shanghai Jiaotong University School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2024-03-12 (Estimated); Primary Completion 2025-06-12 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Whether hypothermia occurs | Generally 1 ~ 3 hours, up to 3 hours can be observed.
  If the patient 's body temperature is lower than 36 °C during this period, it will be determined that the patient has a postoperative hypothermia, and the rewarming measures will be implemented according to the doctor 's advice. If the patient 's body temperature data collected during this period were all greater than or equal to 36 ° C and less than or equal to 37.2 ° C, it was determined that the patient 's body temperature was normal during the postoperative recovery period and no postoperative hypothermia occurred.

IPD SHARING:
Plan to Share IPD: No